CLINICAL TRIAL: NCT04237844
Title: Clinic Features and Long-term Outcome of Different Subgroups of Brochopulmonary Dysplasia in Preterm Infants
Brief Title: Clinic Features and Outcome of BPD (SGBPD)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Wang Jianhui (Other)
Responsible Party: Sponsor-Investigator, Wang Jianhui, Attending doctor, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Other Study IDs: 20191112
Record Dates: First submitted 2019-12-18; First posted 2020-01-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Bronchopulmonary Dysplasia
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- no BPD: In preterm infants(GA<32 weeks and hospital day>14 days )，infants without BPD
- classic BPD: In preterm infants(GA<32 weeks and hospital day>14 days )，There are clinical manifestations and imaging evidence of RDS after birth, the condition is not relieved, FiO2 lasts >25%
- BPD after RDS: In preterm infants(GA<32 weeks and hospital day>14 days )，There are clinical manifestations and imaging evidence of RDS after birth. FiO2<23% within 7 days, and the condition is aggravated to FiO2>25%.
- Delayed BPD: In preterm infants(GA<32 weeks and hospital day>14 days )，There is no RDS performance after birth, FiO2 lasts <25%
- Early, lethal BPD: In preterm infants(GA<32 weeks and hospital day>14 days )，Some infants who die before 36 weeks PMA (between 14 days of postnatal age and 36 weeks) due to persistent parenchymal lung disease and respiratory failure that can not be attributable to other neonatalmorbidities

SUMMARY:
This study described the perinatal high-risk factors and clinical manifestations of the children, and compared the high-risk factors, clinical manifestations and prognosis of BPD among different clinical subtypes by comparison between groups. BPD grading was performed using the 2018 grading standard to compare the distribution of I/II/III BPD among different groups.

ELIGIBILITY:
Inclusion Criteria:

1. Premature infants born at <32 weeks of gestational age;
2. hospitalization time ≥ 14 days;
3. The clinical medical records are complete

Exclusion Criteria:

* • 1) Children with congenital heart, lung malformation and definite chromosomal diseases; 2) children gave up treatment halfway; 3) corrected gestational age 36 weeks before death, the cause of death was confirmed as factors other than respiratory system.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Premature infants born at <32 weeks of gestational age and the hospitalization time ≥ 14 days.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | up to 12 months after birth
  Different subtype of BPD infants against the total BPD infants in corresponding group
Serious respiratory mobidities | up to 18 months after birth
  occurence of at least one of the following: tracheostomy, continued hospitalization for respiratory reasons at or beyond 50weeks PMA; continued oxygen supplement or respiratory support beyond 12months after birth; readmission for respiratory reasons.
Duration of first hospital stay | up to 12 months after birth
  days between admission and first discharge
Days with oxygen supplement | up to 12 months after birth
  days during which the infants were given oxygen
Days of Mechanical Ventilation | up to 12 months after birth
  days during which the infants were given mechanical ventilation

SECONDARY OUTCOMES:
weight | up to 18months after birth
  the measure of infant's length
length | up to 18months after birth
  the measure of infant's weight
head circumference | up to 18months after birth
  the measure of infant's head circumference, which is the occipital-frontal circumference

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shi, Study Director — children's hospital of chongqiong Medical University
Locations (1):
- Children's hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Northway WH Jr, Rosan RC, Porter DY. Pulmonary disease following respirator therapy of hyaline-membrane disease. Bronchopulmonary dysplasia. N Engl J Med. 1967 Feb 16;276(7):357-68. doi: 10.1056/NEJM196702162760701. No abstract available. PMID 5334613
- [Background] Shennan AT, Dunn MS, Ohlsson A, Lennox K, Hoskins EM. Abnormal pulmonary outcomes in premature infants: prediction from oxygen requirement in the neonatal period. Pediatrics. 1988 Oct;82(4):527-32. PMID 3174313
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896
- [Background] Laughon M, Allred EN, Bose C, O'Shea TM, Van Marter LJ, Ehrenkranz RA, Leviton A; ELGAN Study Investigators. Patterns of respiratory disease during the first 2 postnatal weeks in extremely premature infants. Pediatrics. 2009 Apr;123(4):1124-31. doi: 10.1542/peds.2008-0862. PMID 19336371
- [Background] Streubel AH, Donohue PK, Aucott SW. The epidemiology of atypical chronic lung disease in extremely low birth weight infants. J Perinatol. 2008 Feb;28(2):141-8. doi: 10.1038/sj.jp.7211894. Epub 2007 Dec 6. PMID 18059466
- [Background] Panickar J, Scholefield H, Kumar Y, Pilling DW, Subhedar NV. Atypical chronic lung disease in preterm infants. J Perinat Med. 2004;32(2):162-7. doi: 10.1515/JPM.2004.029. PMID 15085893
- [Background] Poindexter BB, Feng R, Schmidt B, Aschner JL, Ballard RA, Hamvas A, Reynolds AM, Shaw PA, Jobe AH; Prematurity and Respiratory Outcomes Program. Comparisons and Limitations of Current Definitions of Bronchopulmonary Dysplasia for the Prematurity and Respiratory Outcomes Program. Ann Am Thorac Soc. 2015 Dec;12(12):1822-30. doi: 10.1513/AnnalsATS.201504-218OC. PMID 26397992
- [Background] Schmidt B. No End to Uncertainty about Inhaled Glucocorticoids in Preterm Infants. N Engl J Med. 2015 Oct 15;373(16):1566-7. doi: 10.1056/NEJMe1509243. No abstract available. PMID 26465990
- [Background] Higgins RD, Jobe AH, Koso-Thomas M, Bancalari E, Viscardi RM, Hartert TV, Ryan RM, Kallapur SG, Steinhorn RH, Konduri GG, Davis SD, Thebaud B, Clyman RI, Collaco JM, Martin CR, Woods JC, Finer NN, Raju TNK. Bronchopulmonary Dysplasia: Executive Summary of a Workshop. J Pediatr. 2018 Jun;197:300-308. doi: 10.1016/j.jpeds.2018.01.043. Epub 2018 Mar 16. No abstract available. PMID 29551318
- [Background] Steinhorn R, Davis JM, Gopel W, Jobe A, Abman S, Laughon M, Bancalari E, Aschner J, Ballard R, Greenough A, Storari L, Thomson M, Ariagno RL, Fabbri L, Turner MA; International Neonatal Consortium. Chronic Pulmonary Insufficiency of Prematurity: Developing Optimal Endpoints for Drug Development. J Pediatr. 2017 Dec;191:15-21.e1. doi: 10.1016/j.jpeds.2017.08.006. No abstract available. PMID 29173299